CLINICAL TRIAL: NCT06891352
Title: Optimization of Chrononutrition to Reduce the Risk of Disease in Shift Workers - The SHIFT Study
Brief Title: Optimization of Chrononutrition to Reduce the Risk of Disease in Shift Workers
Acronym: SHIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salk Institute for Biological Studies (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of San Diego (Other)
Responsible Party: Principal Investigator, Emily N.C. Manoogian, Staff Scientist, Salk Institute for Biological Studies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-0002; 1R01DK139356-01 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Night Shift Work; Time Restricted Eating; Overweight; Obesity
Keywords: Time-Restricted Eating; Night Shift work; Nurses; Nursing Assistants
MeSH Terms: conditions — Intermittent Fasting; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Monitoring (Active Comparator): Log all dietary intake and continue habitual eating patterns.
  Interventions: Behavioral: Dietary Monitoring
- Time-Restricted Eating (TRE) (Experimental): Dietary Monitoring and adherence to a personalized consistent 10-hour time-restricted eating window
  Interventions: Behavioral: Time-Restricted Eating (TRE)
- Time-Restricted Eating with Low-Glycemic Snack (TRE-LGS) (Experimental): Dietary Monitoring and adherence to a modified personalized consistent 10-hour time-restricted eating window a low-glycemic snack provided by the research team to consume during night shifts.
  Interventions: Behavioral: Time-Restricted Eating with a Low-Glycemic Snack (TRE-LGS)

INTERVENTIONS:
Behavioral: Dietary Monitoring — Participants in the group will receive standard advice for a healthy lifestyle, log all food and beverage intake on the myCircadianClock app, and continue their habitual eating patterns.
  Arms: Dietary Monitoring
Behavioral: Time-Restricted Eating (TRE) — Participants in the group will receive standard advice for a healthy lifestyle, log all food and beverage intake on the myCircadianClock app, and adhere to a personalized consistent 10-hour time-restricted eating window.
  Arms: Time-Restricted Eating (TRE)
Behavioral: Time-Restricted Eating with a Low-Glycemic Snack (TRE-LGS) — Participants in the group will receive standard advice for a healthy lifestyle, log all food and beverage intake on the myCircadianClock app, and adhere to a personalized consistent 10-hour time-restricted eating window. On nights that participants work night shifts, they will consume a low-glycemic snack provided by the research team.
  Arms: Time-Restricted Eating with Low-Glycemic Snack (TRE-LGS)

SUMMARY:
In this randomized controlled trial, the investigators will assess the health impacts of optimizing the timing of dietary consumption in nurses and nursing assistants who work night shifts, have a habitual eating window of 14 hours or more, and elevated weight. Participants will be randomized to one of three groups: (1) dietary monitoring, (2) dietary monitoring plus 10-hour daytime time-restricted eating (TRE), or (3) TRE with a low-glycemic snack during night shifts. The study includes a 2-week screening/baseline health assessment, with follow-up health assessments at 3-, 6- (primary outcome), and 12 months.

DETAILED DESCRIPTION:
The purpose of this study is to assess if reducing the number of hours during which participants eat each day, and consolidating dietary intake to the daytime, (with or without a low glycemic snack during night shifts) will help decrease weight and abdominal fat, improve glucose (sugar) regulation, and improve other markers of metabolic and cardiovascular health (i.e. lipid levels, inflammation markers, etc.).

Circadian clocks ("circa" means approximately and "dian" means day) are daily rhythms in physiology and behavior (activity, sleep, eating pattern) that help our body to anticipate and adapt to predictable events in the environment. These rhythms are generated and maintained by biological clocks that are present in the brain and almost every organ of our body. Remarkably, even in the absence of any timing information from a device, our body can keep track of time and thereby help us go to sleep and eat at optimum times. However, our lifestyle and work schedules can lead us to eat, exercise, and sleep at times that the clocks in our body are not prepared for. When these abnormal daily patterns continue for several weeks or years, it can affect our health in many ways including increased body weight, poor sleep, and elevated risk for various chronic diseases. Time-restricted eating (TRE), which restricts all dietary intake to a personalized consistent daily eating window to support circadian rhythms, has been shown to improve cardiometabolic health. However, TRE has not yet been assessed in people who work night shifts.

In this study, the investigators are interested in evaluating the effects of modifying eating patterns on the health of nurses and nursing assistants who work night shifts. Participants will be randomized to (1) dietary monitoring alone, or in combination with, (2) personalized 10-hour TRE (TRE), or (3) personalized 10-hour TRE with a low-glycemic snack provided to consume during night shifts (TRE-LGS). The TRE group will only be allowed water, black coffee, and tea (without any additives such as cream, sweetener including artificial sweeteners), during night shifts. The TRE+LGS group will be provided a low glycemic snack during night shifts.

The study is a year-long including a 2-week screening/baseline assessment, a 6-month guided intervention, and a 6-month self-guided intervention. Health assessments will be taken at screening/baseline, 3 months, 6 months (primary outcome), and 1 year (follow-up). Assessments will include weight (in clinic and at home), blood pressure (in clinic and at home), dietary recall (ASA24), body mass index, blood tests (biomarkers of cardiometabolic health parameters), glycemic regulation (Continuous Glucose Monitors), body composition ( duel energy x-ray absorptiometry, DXA), dietary intake (logged on the myCircadianClock smartphone app), sleep and quality of life questionnaires, and activity, sleep, and wrist temperature (actigraphy watch).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* BMI ≥ 25 kg/m2 (or ≥ 23 kg/m2 for Asian adults)
* Own a smartphone (Apple iOS or Android OS)
* Baseline eating window ≥ 14 h/day
* Night shift nurses and nursing assistants who are working a 12-hour night shift at least 3 days/week.
* Have been doing night shift work for at least 3 months.
* Patients on cardiovascular medications (HMG CoA reductase inhibitors (statins), metformin, lipid-modifying drugs (including over-the-counter drugs such as red yeast rice and fish oil), anti-hypertensive, drugs), are allowed
* If patients have Type 2 Diabetes, they will be included in the study if A1c is less than 9 and they are not on insulin.

Exclusion Criteria:

* Insufficient dietary logging on the mCC app is defined as less than 7 of 14 days of baseline of dietary logging with a minimum of 2 items a day, at least 5 hours apart.
* Type 1 Diabetes or Insulin-dependent Type 2 Diabetes.
* Use of sulfonylurea or insulin within the last 3 months (due to unknown safety with TRE)
* Use of medications that are known to cause weight loss such as SGLT2 inhibitors and GLP1 receptor agonists)
* BMI > 50 kg/m2
* Change in medications that could impact study outcomes within the past 3 months
* Change in weight of >4kg in the past 3 months
* Women who are pregnant, breastfeeding, or are trying to become pregnant during the study period. If a participant becomes pregnant during the study, they will be excluded from continuing the study.
* Systolic BP greater than 160 mmHg and/or diastolic BP greater than 110 mmHg at rest
* Fasting LDL cholesterol greater than 250 mg/dL
* Fasting triglycerides greater than 500g/dL
* Active tobacco abuse or illicit drug use or history of treatment for alcohol abuse in the past 5 years.
* Frequent (more than 4) travel involving a time zone change of more than 3 hours over the 1-year study period
* Prolonged leave from work (a continuous month or longer) during the study
* Active treatment for inflammatory and/or rheumatologic disease
* History of a major adverse cardiovascular event within the past year (acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack)
* Uncontrolled arrhythmia (i.e. rate-controlled atrial fibrillation/atrial flutter are acceptable)
* History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (hypothyroidism on a stable dose of thyroid replacement therapy is allowed).
* History of adrenal disease in the past 5 years
* History of malignancy undergoing active treatment, except non-melanoma skin cancer, in the past 5 years
* History of an eating disorder in the past 5 years
* History of cirrhosis in the past 5 years
* History of stage 4 or 5 chronic kidney disease or dialysis in the past 5 years
* History of HIV/AIDs
* Currently enrolled in weight-loss or weight-management program
* History of surgical intervention for weight management within the past 2 years, or longer if deemed unsafe following review by medical investigators
* Uncontrolled psychiatric disorder including prior hospitalization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-03-03 (Estimated)

PRIMARY OUTCOMES:
Total Body Fat Mass (kg) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Total Body Fat Mass (kg) assessed by DXA

SECONDARY OUTCOMES:
Body weight (kg) in clinic | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Body weight (kg) measured in clinic while participants are wearing a gown that has been weighed.
Body Mass Index | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Body Mass Index (BMI) (kg/m2)
HbA1c (%) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Hemoglobin A1c (%) from fasted blood draw
Intra-Daily Glycemic Variability: CONGA (A.U.) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Continuous Overall Net Glycemic Action (CONGA) assessed via continuous glucose monitor
Inter-Daily Glycemic Variability: MODD (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Mean of Daily Differences (MODD) assessed via continuous glucose monitor
Glycemic Variability: MAGE (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Mean Amplitude of Glycemic Excursions (MAGE) assessed by continuous glucose monitor
Mean Glucose (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Mean Glucose assessed by continuous glucose monitor
Fasting Glucose (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Blood glucose assessed from a fasted blood draw
Fasting Insulin (uIU/mL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Blood insulin assessed from a fasted blood draw
Blood Pressure (mmHg) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Systolic and Diastolic Blood Pressure taken in clinic.
Blood Pressure (mmHg)_at home measurements | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Systolic and Diastolic blood pressure taken at home. Measurements are taken twice (one measurement on a work day and one on an off day) during the 2 week assessment periods. Each day measurements will be taken 3 times throughout the day. Averages for work days and off days will be reported for each time point. Averages at each time point will be reported.
Direct LDL Cholesterol (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Direct LDL cholesterol from fasted blood draw
Non-HDL Cholesterol (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Non-HDL cholesterol from fasted blood draw

OTHER OUTCOMES:
Lean Mass (g) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Whole body lean mass (g) assessed by DXA scan
Percent Body Fat (%) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Whole body percent Body Fat (%) assessed by DXA scan
Visceral Adipose Tissue Mass (g) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Whole body Visceral Adipose Tissue Mass (g) assessed by DXA scan
Body Weight (kg) at home | From enrollment to the end of the intervention at 1 year.
  Participants will weigh themselves every 2 weeks at home on study provided scales in the morning.
Blood Glucose Time in Range (%) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Time in range (%) from continuous glucose monitor.
Glycemic Management Indicator (%) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Glycemic Management Indicator (GMI, %), an estimate of A1c, from continuous glucose monitor.
Triglycerides (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Triglycerides (mg/dL) from fasted blood draw.
Total Cholesterol (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Total cholesterol (mg/dL) from fasted blood draw.
HDL-cholesterol (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  HDL-cholesterol (mg/dL) from fasted blood draw.
hs-CRP (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  hs-CRP (mg/dL) from a fasted blood draw.
LDL Particle number (nmol/L) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  LDL Particle number (nmol/L) assessed by NMR lipoprotein profiles from a fasted blood draw.
Apo A (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Apo A (mg/dL) assessed by NMR lipoprotein profiles from a fasted blood draw.
Apo B (mg/dL) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Apo B (mg/dL) assessed by NMR lipoprotein profiles from a fasted blood draw.
Apo A/B ratio | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Apo A/B ratio assessed by NMR lipoprotein profiles from a fasted blood draw.
Very Low Density Lipoprotein (VLDL) Size (nm) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  VLDL size (nm) assessed by NMR lipoprotein profiles from a fasted blood draw.
HDL Particle number (umol/L) | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  HDL Particle number (umol/L) assessed by NMR lipoprotein profiles from a fasted blood draw.
Quality of Life Assessment | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Short-Form 36 (SF-36) Survey. Scores range from 0-100 (an average of all questions which each have a 0-100 scale), with 100 indicating better physical and emotional health.
Sleep Duration | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Average total daily sleep duration assessed by actigraphy watch
Pittsburgh Sleep Quality Index | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Pittsburgh Sleep Quality Index (PSQI). Each item is scored on a 0-3 scale with a total score of 0-21. A lower score indicates better sleep.
Epworth Sleepiness Scale | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Epworth Sleepiness Scale (ESS). Scored from 0-24. A lower score indicates less sleepiness.
Chronotype | Baseline, 3 month, 6 month (primary), and 12 month (follow-up)
  Munich Chronotype Questionnaire (MCTQ) Shiftwork estimates an individuals chronotype.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Manoogian, Ph.D., Principal Investigator — Salk Institute for Biological Studies
Locations (1):
- University of California San Diego Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will report deidentified individual participant data for outcomes that are reported in scientific publications (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 1 month of publication with no set end date (minimum of 5 years).
Access Criteria: Data will be available to anyone who wants to access it through a data depository that will be disclosed at the time of publication.